CLINICAL TRIAL: NCT02725021
Title: Education Against Tobacco: Medical-student-delivered Smoking Prevention Programme for Secondary Schools in Brazil - Randomized Trial
Brief Title: Education Against Tobacco Randomized Trial in Brazil
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Giessen (Other)
Responsible Party: Principal Investigator, Titus J. Brinker, Principal Investigator, University of Giessen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EATBrazil
Record Dates: First submitted 2016-03-13; First posted 2016-03-31 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2016-04

CONDITIONS: Tobacco Prevention
Keywords: tobacco prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): The intervention group receives a school-based module taking about two hours delivered by medical students in the schools.
  Interventions: Behavioral: Education Against Tobacco school-based intervention by medical students
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Education Against Tobacco school-based intervention by medical students
  Arms: Intervention group

SUMMARY:
A two armed randomized trial is evaluating the effect of the medical-student-delivered school-based intervention Education Against Tobacco on the smoking behavior of adolescents in 7-11th grade of secondary school. The primary endpoint is the change in smoking prevalence between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Visiting grades 7-11 of a regular public secondary school in Brazil.

Exclusion Criteria:

* Not fulfilling inclusion criteria.

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1500 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-02 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Smoking prevalence measured via questionnaire. | 12 months follow-up

SECONDARY OUTCOMES:
Smoking onset: Difference in the number of new smokers at 12 months of follow-up who were not present at baseline | Baseline and 12 months
Difference in the number of new non-smokers at 12 months of follow-up who were smoking at baseline | Baseline and 12 months
Relevant differences due to the theory of planned behaviour between the two groups measured via questionnaire. | Difference in attitude towards smoking between the two groups at 12 months follow-up measured via questionnaires.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lisboa OC, Bernardes-Souza B, Xavier LEF, Almeida MR, Correa PCRP, Brinker TJ. A Smoking Prevention Program Delivered by Medical Students to Secondary Schools in Brazil Called "Education Against Tobacco": Randomized Controlled Trial. J Med Internet Res. 2019 Feb 21;21(2):e12854. doi: 10.2196/12854. PMID 30789347
- [Derived] Xavier LE, Bernardes-Souza B, Lisboa OC, Seeger W, Groneberg DA, Tran TA, Fries FN, Correa PC, Brinker TJ. A Medical Student-Delivered Smoking Prevention Program, Education Against Tobacco, for Secondary Schools in Brazil: Study Protocol for a Randomized Trial. JMIR Res Protoc. 2017 Jan 30;6(1):e16. doi: 10.2196/resprot.7134. PMID 28137703